CLINICAL TRIAL: NCT01432119
Title: Phase I Trial of Cetuximab and Erlotinib (EGFR Inhibitors) and SIR-Spheres (Yttrium Microspheres) in Patients With Advanced Malignancies and Liver Metastases
Brief Title: Phase 1 Trial With SIR-Spheres and Cetuximab +/- Erlotinib
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0552
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Advanced Malignancies; Liver Metastases; SIR-Spheres; Selective internal radiation; Yttrium-90; Cetuximab; C225; Erbitux; Erlotinib; Erlotinib Hydrochloride; Tarceva; OSI-774
MeSH Terms: interventions — Cetuximab; Erlotinib Hydrochloride; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 SIR-Spheres + Cetuximab (Experimental): Arm 1: SIR-Spheres with yttrium-90 attached and cetuximab. SIR-Spheres Day 1 of Cycle 1; Cetuximab start 200 mg/m2 by vein (IV) Weeks 2-4 of Cycle 1, then weekly Cycles 2+. 28-day Cycles. Nuclear medicine "break-through" scan performed within 29 days before receiving SIR-Spheres. The results of this test will be used to determine if a full or partial dose of SIR-Spheres with yttrium-90 microspheres will be delivered.
  Interventions: Device: SIR-Spheres; Drug: Cetuximab; Procedure: Break-Through Scan
- Arm 2 SIR-Spheres + Cetuximab + Erlotinib. (Experimental): Arm 2: SIR-Spheres with yttrium-90 attached, cetuximab, and erlotinib. Physicians will assign patients to Arm 1 or Arm 2 based on their discretion. SIR-Spheres on Day 1 of Cycle 1; Cetuximab start 200 mg/m2 by vein (IV) Weeks 2-4 of Cycle 1, then weekly Cycles 2+. 28-day Cycles. Erlotinib start 100 mg by mouth daily starting with Cycle 2. 28-day Cycles. Nuclear medicine "break-through" scan performed within 29 days before receiving SIR-Spheres. The results of this test will be used to determine if a full or partial dose of SIR-Spheres with yttrium-90 microspheres will be delivered.
  Interventions: Device: SIR-Spheres; Drug: Cetuximab; Drug: Erlotinib; Procedure: Break-Through Scan

INTERVENTIONS:
Device: SIR-Spheres — 100% full dose SIR-Spheres on Day 1 of Cycle 1. SIR-Spheres with yttrium-90 microspheres will be given through a catheter in a vein in the groin.
Drug: Cetuximab — Starting Dose: 200 mg/m2 by vein weekly. During Cycle 1, patients will receive cetuximab during Weeks 2-4. In Cycles 2 and beyond, patients will receive cetuximab weekly.
  Other Names: C225; Erbitux
Drug: Erlotinib — Starting dose: 100 mg by mouth daily. Erlotinib will be given starting with Cycle 2 at 100 mg by mouth daily. If tolerated, the dose will be increased to 150 mg by mouth daily in Cycle 3.
  Other Names: Erlotinib Hydrochloride; OSI-774; Tarceva
  Arms: Arm 2 SIR-Spheres + Cetuximab + Erlotinib.
Procedure: Break-Through Scan — Nuclear medicine "break-through" scan performed within 29 days before receiving SIR-Spheres. The results of this test will be used to determine if a full or partial dose of SIR-Spheres with yttrium-90 microspheres will be delivered.
  Other Names: x-ray

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of selective internal radiation (SIR)-Spheres with yttrium-90 attached and cetuximab. Some participants will also take erlotinib with this combination.

Yttrium-90 microspheres are designed to treat cancer that has spread to the liver. SIR-Spheres are designed to deliver the radiation directly to the liver. This radiation may cause the tumor cells to die.

Cetuximab and erlotinib are drugs that are designed to block the epidermal growth factor receptor (EGFR). EGFR is a protein that helps cancer cells grow. Blocking the EGFR may stop tumors from growing.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, your doctor will decide which group you will be in based on your medical history.

* Group 1 will receive SIR-Spheres with yttrium-90 attached and cetuximab.
* Group 2 will receive SIR-Spheres with yttrium-90 attached, cetuximab, and erlotinib.

Once it is decided which combination you will receive, you will be assigned to a dose level of cetuximab based on when you join the study. Up to 3 dose levels of cetuximab will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable doses of the combinations are found.

All study participants will receive a dose level of the SIR-Spheres with yttrium-90 attached based on the results of the "break-through" scan (described below).

If you are assigned to Group 2, you will also receive erlotinib. If you are tolerating erlotinib well after 1 cycle, you may begin receiving a higher dose of erlotinib in Cycle 3 and beyond.

Break-through Scan:

You will have a "break-through" scan within 29 days before receiving the SIR-Spheres with yttrium-90 microspheres. This scan will measure the supply of blood in your lungs and will also be used to check your liver. For this test, a small amount of radioactive material will be injected into your liver and images will be taken to see how the material moves through your lungs and liver. The radioactive material will be given through a catheter in a vein in your groin. A catheter is a sterile, flexible tube that will be placed through your groin artery into the artery leading to your liver while you are under local anesthesia. Your doctor will explain this procedure to you in more detail.

The results of this test will be used to determine if you will receive a full or partial dose of SIR-Spheres with yttrium-90 microspheres.

Radiation and Study Drug Administration:

Each study cycle is 28 days.

You will receive the SIR-Spheres with yttrium-90 microspheres on Day 1 of Cycle 1 only. Before you receive the SIR-Spheres with Yttrium-90 microspheres, you will receive sedative drugs by vein to put you to sleep. SIR-Spheres with yttrium-90 microspheres will then be given to you through a catheter in a vein in your groin.

After you are given the yttrium-90 microspheres, the catheter will be removed and pressure will be applied to your groin to stop any bleeding. You will then be monitored for 6 hours to check for any side effects. If needed, you will be given pain medication after the infusion. Your study doctor will decide which pain medications to give you.

Cetuximab will be given by vein 1 time each week during Weeks 2-4 of Cycle 1, and then 1 time every week for Cycles 2 and beyond. The first time you receive cetuximab, it will be given over 2 hours. Every time you receive cetuximab after that, it will be given over 1 hour.

If you are assigned to receive erlotinib, you will take it by mouth 1 time each day starting on Day 1 of Cycle 2. You should take it at the same time each day . You should take it on an empty stomach either 1 hour before or 2 hours after eating. The study staff will give you more instructions for taking erlotinib.

Study Visits:

On Day 1 of Cycle 1:

* Before you receive the SIR-Spheres with yttrium-90 microspheres, your blood vessels will be checked. For this test, you will receive an x-ray dye through the catheter that will help the study staff look at the arteries leading to your liver and surrounding areas.
* You will have a physical exam and your medical history will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

During Weeks 2 and 4 of Cycle 1:

* You will have a physical exam and your medical history will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Every 8 weeks, you will have an x-ray, CT scan, MRI scan, and/or PET/CT scan to check the status of the disease.

About every 4 weeks starting at the beginning of Cycle 2:

* You will have a physical exam and your medical history will be recorded
* Blood (about 2 teaspoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test if you are able to become pregnant.

Length of Study:

You receive the study drugs for as long as you are benefitting. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. SIR-Spheres are FDA-approved and commercially available to treat metastatic colorectal cancer that has spread to the liver. Yttrium-90 microspheres are FDA-approved for hepatic arterial therapy and the treatment of liver metastases. Cetuximab is FDA-approved and commercially available to treat head and neck and colorectal cancer. Erlotinib is FDA-approved and commercially available to treat non-small cell lung cancer (NSCLC) and pancreatic cancer. The use of this combination to treat advanced cancer is investigational.

Up to 136 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer in the liver, with measureable or evaluable disease, that is refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months
2. Patients must be >/= 3 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery. Patients may have received palliative localized radiation immediately before or during treatment providing radiation is not delivered to the only site of disease being treated under this protocol
3. ECOG performance status </= 3.
4. Patients must have organ and marrow function defined as: • Absolute neutrophil count >/= 500/mL; • Platelets >/=50,000/mL; creatinine </= 2 X ULN; • Total bilirubin </= 2.0; ALT(SGPT) </= 5 X ULN
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence).
6. Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients who have had hepatic external beam radiotherapy.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to SIR-Spheres, cetuximab, or erlotinib.
4. Patients with colorectal cancer with known kRAS mutation
5. Hepatic arterial anatomy that would prevent catheterization and the administration of SIR-Spheres into the liver.
6. Greater than 20% arterio-venous shunting of SIR-Spheres to the lungs estimated from a Technetium-99m-macro-aggregated albumin (99mTc-MAA) nuclear medicine break-through scan
7. Contraindication to angiography and selective visceral catheterization: History of severe allergy or intolerance to any contract media, or atropine. Bleeding diathesis, not correctable by usual forms of therapy that would include medical coagulopathy but not limited to the administration of blood products.
8. Utilization of capecitabine for the 6 weeks preceding SIR-Spheres therapy and indefinitely following SIR-Spheres therapy as per manufacturer's recommendations due to the increased risk of radiation hepatitis.
9. Evidence of ascites, biopsy proven cirrhosis, or portal hypertension suggested by the presence of characteristic imaging features on cross-sectional imaging or esophageal varicosities, demonstrated on endoscopy or barium swallow. A diagnostic study to rule out the presence of portal hypertension will not be required unless the findings on cross sectional imaging are suggestive, but not confirmatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 8 weeks
  Maximum tolerated dose (MTD) is defined as the highest dose studied in which the incidence of dose limiting toxicities (DLT) was less than 33% of treated population.

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org